CLINICAL TRIAL: NCT03826628
Title: A Phase 2/3, Multi-Center, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Dose-Response Comparison of the Efficacy and Safety of a Topical Rapamycin Cream for the Treatment of Facial Angiofibromas (FA) Associated With Tuberous Sclerosis Complex (TSC) in Patients 6 Years of Age and Over
Brief Title: Dose-Ranging Efficacy and Safety Study of Topical Rapamycin Cream for Facial Angiofibroma Associated With Tuberous Sclerosis Complex
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dermatology Specialties Limited Partnership (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSLP-01
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-07

CONDITIONS: Facial Angiofibroma; Tuberous Sclerosis
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5% Rapamycin cream, topical (Experimental): Rapamycin cream topical, 0.5% w/w, applied once daily before bed on affected area for 26 weeks
  Interventions: Drug: rapamycin
- 1.0% Rapamycin cream, topical (Experimental): Rapamycin cream topical, 0.5% w/w, applied once daily before bed on affected area for 26 weeks
  Interventions: Drug: rapamycin
- Placebo (Placebo Comparator): Placebo cream topical, applied once daily before bed on affected area for 26 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rapamycin — Apply to the affected area once a day, approximately half an hour before retiring for bed in the evening, for 26 weeks
  Other Names: sirolimus
  Arms: 0.5% Rapamycin cream, topical; 1.0% Rapamycin cream, topical
Drug: placebo — Apply to the affected area once a day, approximately half an hour before retiring for bed in the evening, for 26 weeks
  Arms: Placebo

SUMMARY:
The study aims to compare the safety and efficacy of two different strengths of Rapamycin cream, topical and placebo over 26 weeks in the treatment of facial angiofibroma (FA) associated with Tuberous Sclerosis Complex (TSC).

DETAILED DESCRIPTION:
Topical rapamycin has previously been used to treat FA associated with TSC, reducing erythema, papule size, while flattening lesions and improving skin texture. Topical rapamycin has been reported to be well tolerated.

The efficacy and safety of a topical rapamycin cream at two strengths (0.5% and 1.0%) will be assessed during a 26 week double-blind treatment phase with assessments made at clinical visits at baseline, 2, 8, 14, 20 and 26 weeks, and at follow-up (4 weeks after the last dose of study drug).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 6 years and ≤ 65 years on the day informed consent is obtained
2. Patients diagnosed with TSC based on the clinical diagnostic criteria of International Tuberous Sclerosis Complex Consensus Conference 2012 and presenting visible facial angiofibroma
3. An FA severity score of 2 or 3 on the IGA scale
4. Patients or their legal representatives capable of understanding the explanation of the clinical trial and who give written informed consent for participation
5. Patients or their legal representatives able to maintain patient diaries following the instructions of the investigator or sub-investigator

Exclusion Criteria:

1. Patients who cannot carry out the treatment plan or follow-up assessment
2. Patients with serious skin lesions such as erosions or ulcers
3. Patients with known hypersensitivity to any component of the study product
4. Patients who have received rapamycin/sirolimus, everolimus, or temsirolimus within 3 months of enrolment
5. Patients who received laser therapy or surgical therapy within 6 months prior to trial enrolment
6. Patients who participated in any other clinical trial within 3 months prior to the day of enrolment
7. Patients judged unsuitable for this clinical trial by the investigator or sub-investigator
8. Pregnant or lactating females
9. Sexually active females of childbearing potential not using adequate contraception and sexually active males not using adequate contraception
10. Patients with immune dysfunction or receiving any form of immunosuppression
11. Patients with severe FA, with a score of 4 on the IGA scale
12. Patients with an FA severity score of less than 2 on the IGA scale

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Stanescu, Study Director — Dermatology Specialties Limited Partnership
Locations (17):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - All Children's Research Institute, St. Petersburg, Florida
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia, Charlottesville, Virginia
- Children's Health Queensland, Brisbane, Queensland, Australia
- Fakultni nemocnice Brno, Brno, Czechia
- Hungary (2):
  - Bethesda Children's Hospital of the Hungarian Reformed Church, Budapest
  - University of Pécs, Pécs
- Canterbury District Health Board, Christchurch, Canterbury, New Zealand
- Serbia (2):
  - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade
  - Clinical Center of Serbia, Belgrade
- Narodný ústav detských chorȏb, Bratislava, Slovakia
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clínica Universidad de Navarra, Madrid
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is not planned to be shared with other researchers

REFERENCES:
- [Result] Aitken P, Stanescu I, Boddington L, Mahon C, Fogarasi A, Liao YH, Ivars M, Moreno-Artero E, Trauner D, DeRoos ST, Jancic J, Nikolic M, Balazova P, Price HN, Hadzsiev K, Riney K, Stapleton S, Tollefson MM, Bauer D, Pinkova B, Atkinson H. A novel rapamycin cream formulation improves facial angiofibromas associated with tuberous sclerosis complex: a double-blind randomized placebo-controlled trial. Br J Dermatol. 2023 Oct 25;189(5):520-530. doi: 10.1093/bjd/ljad243. PMID 37463422

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.0% Rapamycin Cream, Topical: Rapamycin cream topical, 1.0% w/w, applied once daily before bed on affected area for 26 weeks
  rapamycin: Apply to the affected area once a day, approximately half an hour before retiring for bed in the evening, for 26 weeks
Period: Overall Study
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Started | 36 | 33 | 38
Completed | 32 | 31 | 35
Not Completed | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo | Total
Number analyzed (Participants) | 36 | 33 | 38 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (15) | 25.5 (15) | 26.3 (13.8) | 26.6 (14.5)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 6-11 years | 6 | 4 | 6 | 16
  Age group: 12-17 years | 5 | 8 | 7 | 20
  Age group: 18-65 years | 25 | 21 | 25 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 23 | 58
  Male | 15 | 19 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 4 | 13
  Not Hispanic or Latino | 31 | 29 | 34 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 7 | 5 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 28 | 26 | 30 | 84
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Study Site [Count of Participants; unit: Participants]
  Site #00 - ACRI Johns Hopkins | 0 | 0 | 2 | 2
  Site #01 - University Hospital Brno | 1 | 0 | 0 | 1
  Site #02 - Children's Health Queensland | 1 | 1 | 0 | 2
  Site #03 - Christchurch Hospital | 2 | 2 | 3 | 7
  Site #04 - University of Navarra | 4 | 4 | 3 | 11
  Site #05 - Mayo Clinic | 1 | 0 | 1 | 2
  Site #06 - Phoenix Children's Hospital | 2 | 2 | 1 | 5
  Site #07 - Spectrum Health, Michigan | 3 | 3 | 3 | 9
  Site #08 - University of California, San Diego | 3 | 4 | 2 | 9
  Site #09 - University of Virginia | 1 | 0 | 1 | 2
  Site #10 - University of Pecs | 1 | 1 | 2 | 4
  Site #11 - Slovakia National Institute of Children's Diseases | 3 | 2 | 2 | 7
  Site #12 - Bethesda Children's Hospital | 5 | 4 | 7 | 16
  Site #13 - University of Szeged | 0 | 0 | 0 | 0
  Site #14 - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade | 2 | 3 | 3 | 8
  Site #15 - Clinical Center of Serbia | 2 | 2 | 3 | 7
  Site #16 - National Taiwan University | 5 | 5 | 5 | 15
Height [Mean (Standard Deviation); unit: centimeters] | 164 (17) | 165 (16) | 161 (17) | 163 (17)
Weight [Mean (Standard Deviation); unit: kilograms] | 68.1 (22.8) | 68.9 (24.3) | 68.4 (25.8) | 68.5 (24.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (5.6) | 24.8 (6.6) | 25.4 (6.4) | 25 (6.2)
Rapamycin concentration [Count of Participants; unit: Participants]
  Below limit of detection | 36 | 33 | 38 | 107
  Above limit of detection | 0 | 0 | 0 | 0
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — The Investigator's Global Assessment (IGA) measures the severity of facial angiofibroma, with scores between 0 (clear) and 4 (severe).
  0 = Clear
  1. = Almost Clear
  2. = Mild
  3. = Moderate
  4. = Severe
  Participants
    2 - Mild | 13 | 16 | 19 | 48
    3 - Moderate | 23 | 17 | 19 | 59
Facial Angiofibroma Severity Index (FASI) [Count of Participants; unit: Participants] — Facial Angiofibroma Severity Index (FASI) grades lesions according to their erythema, size and extent. Scores range between 2 and 9. Scores are summed from the following measures:
  Erythema Skin color 0 Light Red 1 Red 2 Dark Red/purple 3 Size None 0 Small (< 5mm) 1 Large (> 5mm) 2 Confluent 3 Extension <50 % cheek surface 2 >50% cheek surface 3
  Participants
    4 | 7 | 5 | 6 | 18
    5 | 12 | 13 | 16 | 41
    6 | 8 | 6 | 8 | 22
    7 | 6 | 5 | 5 | 16
    8 | 2 | 3 | 3 | 8
    9 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Obtaining Successful Treatment
Description: Success on the Investigator Global Assessment (IGA) scale is defined as clear or almost clear with an improvement of at least two grades from baseline. IGA scores range from 0-4:
  0=Clear
  1. Almost Clear
  2. Mild
  3. Moderate
  4. Severe
Time Frame: After 26 weeks treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Participants | 4 | 3 | 2

2. Secondary Outcome: Time to Treatment Success
Description: The time elapsed from the first dose to the time of treatment success, according to the Investigator's Global Assessment (IGA) scale. The total time of treatment was 26 weeks, although Covid-19 visit delays led to an extension of up to 2 weeks (28 weeks total) for some patients. Success on the Investigator Global Assessment (IGA) scale is defined as clear or almost clear with an improvement of at least two grades from baseline. IGA scores range from 0-4:
  0=Clear
  1. Almost Clear
  2. Mild
  3. Moderate
  4. Severe
Time Frame: From first dose to 26 weeks (± 2 weeks)
Measure: Mean (Standard Error); unit: weeks
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
weeks | 25.89 (0.7) | 26.71 (0.28) | 19.7 (0.22)

3. Secondary Outcome: Change From Baseline in Investigator's Global Assessment
Description: The change in grading on the Investigator's Global Assessment (IGA) scale from baseline.
  IGA scores range from 0-4:
  0=Clear
  1. Almost Clear
  2. Mild
  3. Moderate
  4. Severe
Time Frame: At baseline and after 26 weeks treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Participants
  -2 | 4 | 3 | 2
  -1 | 16 | 17 | 7
  0 | 15 | 13 | 28
  +1 | 0 | 0 | 1
  Missing | 1 | 0 | 0

4. Secondary Outcome: Change From Baseline in Facial Angiofibroma Severity Index (FASI)
Description: The change in grading on the Facial Angiofibroma Severity Index (FASI) from baseline. FASI grades lesions according to their erythema, size and extent by summing the scores of each category. The final FASI scores range from (mild) 2-9 (severe).
  Erythema Skin color 0 Light Red 1 Red 2 Dark Red/purple 3 Size None 0 Small (< 5mm) 1 Large (> 5mm) 2 Confluent 3 Extension <50 % cheek surface 2 >50% cheek surface 3
Time Frame: At baseline and after 26 weeks treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Participants
  -5 | 1 | 1 | 0
  -4 | 1 | 3 | 1
  -3 | 6 | 3 | 1
  -2 | 10 | 9 | 3
  -1 | 10 | 13 | 17
  0 | 7 | 4 | 14
  +1 | 0 | 0 | 1
  +2 | 0 | 0 | 1
  Missing | 1 | 0 | 0

5. Secondary Outcome: Subjective (Participant or Parent/Caregiver) Percentage Change Rating Scale
Description: Percentage change in facial angiofibroma since beginning treatment, as assessed by the participant or parent/caregiver. A large value indicates most improvement to facial angiofibroma (minimum=0, maximum=100). This was a single assessment time-point, where the participant or parent/caregiver estimated the percentage change in the facial angiofibroma lesion appearance from their perspective since baseline.
Time Frame: After 26 weeks treatment
Measure: Mean (Standard Error); unit: Percentage Change
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Percentage Change | 57.06 (4.36) | 54.06 (5.21) | 30.84 (3.89)

6. Secondary Outcome: Objective (Clinician) Percentage Change Rating Scale
Description: Percentage improvement in facial angiofibroma since beginning treatment, as assessed by the clinician. A large value indicates most improvement to facial angiofibroma (minimum=0, maximum=100). This was a single assessment time-point, where clinicians estimated the percentage change in the facial angiofibroma lesion appearance from their perspective since baseline.
Time Frame: After 26 weeks treatment
Measure: Mean (Standard Error); unit: Percentage Change
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Percentage Change | 47.83 (3.88) | 49.39 (5.22) | 20.76 (4.05)

7. Secondary Outcome: Categorical Change in Facial Angiofibroma
Description: Change in facial angiofibroma since beginning treatment on a 5-point scale, as assessed by the participant or parent/caregiver. This was a single assessment time-point, where the participant or parent/caregiver evaluated the change in the facial angiofibroma lesion appearance from their perspective since baseline.
Time Frame: After 26 weeks treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
Number analyzed (Participants) | 36 | 33 | 38
Participants
  -1 - Worse | 1 | 0 | 0
  0 - No Difference | 0 | 1 | 12
  +1 - Slightly Better | 2 | 7 | 11
  +2 - Moderately Better | 13 | 7 | 9
  +3 - Significantly Better | 16 | 13 | 4
  Missing | 4 | 5 | 2

ADVERSE EVENTS:
Time Frame: 30 weeks
Description: Adverse events were collected during each clinical visit and follow-up visit. Patients or their parents/guardians were questioned by the investigator regarding any adverse events experienced since the previous clinical visit.
Arm/Group | 0.5% Rapamycin Cream, Topical | 1.0% Rapamycin Cream, Topical | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/33 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/36 | 2/33 | 2/38
Other Adverse Events (participants affected / at risk) | 29/36 | 27/33 | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% Rapamycin Cream, Topical (N=36) | 1.0% Rapamycin Cream, Topical (N=33) | Placebo (N=38)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Constipation, nausea, malnutrition, diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney bleeding (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Collapsed lung (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% Rapamycin Cream, Topical (N=36) | 1.0% Rapamycin Cream, Topical (N=33) | Placebo (N=38)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 13 (15) | 6 (7) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 12 (13) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (7) | 4 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (2)
Skin tightness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 4 (5) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (2) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (3)
Haemorrhage (Vascular disorders) | 2 (2) | 3 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 2 (4)

LIMITATIONS AND CAVEATS:
Covid-19 pandemic halted recruitment, leading to a smaller number of patients recruited than intended (107/120).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03826628/Prot_SAP_000.pdf